CLINICAL TRIAL: NCT00676286
Title: Biological Investigations in Active Surveillance (BIAS) IGAR 2008 I 19
Brief Title: Biological Investigations in Active Surveillance (BIAS) IGAR 2008 I 19 in Prostate Cancer Using High Field MRI (3 Tesla), PET, and Biomarkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GU-24152
Record Dates: First submitted 2008-05-12; First posted 2008-05-13 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer active surveillance; 3 Tesla MR biological imaging in prostate cancer; tumor gene re-arrangements in prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gene Rearrangement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: 3T MR Imaging — 3TR Imaging
Procedure: C-Choline PET Scanning — C-Choline PET Scanning
Procedure: Gene Rearrangement — Gene Rearrangement

SUMMARY:
This study will use high field MRI (3 Tesla), PET and biomarker to follow prostate cancers and determine if these tests can detect cancers that become aggressive.

DETAILED DESCRIPTION:
This study may lead to the identification of additional investigations that can monitor for signs of disease progression in active surveillance protocols. This can directly benefit patients by providing them with greater confidence that their disease is being accurately monitored. In addition, this study may be beneficial to the general management of prostate cancers by adding to our knowledge of these investigations characterizing prostate cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Registration must occur within 16 weeks of last biopsy
* History and physical exam (including DRE) within 8 weeks prior to registration
* Patients must have indolent prostate cancer including all of the following: Low risk prostate cancer, less or equal to 50 % of core biopsies involved with disease, and less or equal to three biopsies involved with disease
* Patients must have a minimum of six biopsies (sextant) at registration
* PSA test within 8 weeks registration
* Creatinine level below 100 umol/L within 8 weeks of registration
* Patients must have no contraindications to MRI scans
* No history of previous malignancies except non-melanoma skin tumors or other malignancies with a greater than 5 year life expectancy
* Patients must be reliable for follow up

Exclusion Criteria:

* Patient does not have histologically-proven adenocarcinoma of the prostate
* Last biopsy greater than 16 weeks prior to registration
* History and physical exam (including DRE) greater that 8 weeks prior to registration
* Patient does not have indolent disease
* Patient has less than six sextant biopsies at registration
* PSA test done greater than 8 weeks from registration
* Creatinine level greater than 100 umol/L within 8 weeks of registration
* Contraindications to MRI scans
* History of previous malignancies other than non-melanoma skin tumors or other malignancies with a greater than 5 year life expectancy
* Patients that are not reliable for follow up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Primary objective to determine if we can accrue patients to this study in a timely manner. | 2 years

SECONDARY OUTCOMES:
Patient compliance | Patients followed for 5 years from baseline
Optimal imaging parameters to characterize prostate cancers | patients followed for 5 years from baseline
feasibility of detecting gene arrangements in prostate biopsies | patients followed for 5 years from baseline
Incidence of patients developing progressive prostate cancer warranting definitive treatment in an active surveillance protocol | patients followe for 5 years from baseline
The natural history of prostate cancer with these investigations | patients followed for 5 years from baseline
The sensitivity and specificity of these investigation in detecting prostate cancer | patients followed for 5 years from baseline
The sensitivity and specificity of these investigations in differentiating indolent prostate cancer from aggressive disease | patients followed for 5 years from baseline
The sensitivity and specificity of these investigations in detecting high grade disease, extracapsular disease and extraprostatic disease and disease progression | patients followed for 5 years from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nawaid Usmani, MD, FRCPC, Study Chair — Cross Cancer Institute; Nawaid Usmani, MD, FRCPC, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada